CLINICAL TRIAL: NCT06010706
Title: Efficacy of Supervised Manual Physical Therapy Exercise for Ankle Disability After Motor Vehicle Accidents, Randomized Controlled Trial.
Brief Title: Supervised Manual Physical Therapy Exercise for Ankle Disability After Motor Vehicle Accidents.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jouf University (Other)
Responsible Party: Principal Investigator, Mosaad, Principal investigator, PhD , Department of physical therapy and Health Rehabilitation, College of applied medical sciences, Jouf University., Jouf University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 123456
Record Dates: First submitted 2023-08-20; First posted 2023-08-24 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Ankle Deformity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supervised Manual Physical Therapy Program (Experimental): Participants will receive a supervised physical therapy program including: mobilizing exercises, stretching exercises, and strengthening exercises. 3 sessions a week for eight consecutive weeks.
  Interventions: Other: Supervised physical therapy manual exercise program.
- Home based exercise program: (Active Comparator): Patients at the control group will receive instruction for home based exercise program of physical therapy exercise. The home program primarily consisted of exercises targeting deficits in joint ROM, muscle flexibility and strength, and balance. The home-based program will include stretching, ROM and strengthening exercises
  Interventions: Other: Stretching exercise, ROM, Strengthening exercises.

INTERVENTIONS:
Other: Supervised physical therapy manual exercise program. — 1. Mobilization Techniques :
     The joint mobilization technique will be the anterior-posterior glide of the talus. The participant will be positioned in supine or long sitting.
  2. Stretching Exercise:
     Passive stretching with therapist assistance was used for ankle dorsiflexion with the knee both flexed and extended. Force during passive stretching was modified to patient tolerance. Each participant flexed the knee slightly while standing on a 10° incline board. The participant was asked to slightly flex both knees until a stretch was felt in the calf muscle.
  3. Strengthening Exercise:
  The resistance training protocol will be based on the progressive resistance training principle and was a modification of the protocol used by Frontera et al [10] in older men. Plantar-flexion resistance training will be performed on a customized hydraulic apparatus, which provide a constant resistance over the entire ROM and allow for concentric as well as eccentric.
  Arms: Supervised Manual Physical Therapy Program
Other: Stretching exercise, ROM, Strengthening exercises. — Patients at the control group will receive instruction for home based exercise program of physical therapy exercise. The home program primarily consisted of exercises targeting deficits in joint ROM, muscle flexibility and strength, and balance.
  Arms: Home based exercise program:

SUMMARY:
Every year more than 50 million people worldwide are injured due to RTAs which in turn makes it one of the leading causes of disability. During automobile collisions, the lower limbs are the most commonly injured region of the human body. Ankle injuries can be particularly long-lasting, resulting in excessive medical costs, inability to work, and serious psychological distress. Physiotherapists often contribute to the rehabilitation of ankle fractures, which typically starts soon after the period of immobilization. Joint mobilization led to increased ankle movement, improved gait patterns, reduced pain and the number of treatment sessions required, and hastened return to activities when compared with the usual rest, ice, compression, and elevation protocol.

DETAILED DESCRIPTION:
Participants will be assigned into two groups:

1. Study group will receive a Supervised physical therapy exercise program in the form of Mobilization exercise, Stretching exercise, and Strengthening exercise.
2. Control group will receive a Home-based exercise program of Stretching exercises, strengthening exercises and ROM exercises.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Stable ankle fractures after motor vehicle accidents involving the distal tibia, distal fibula, or talus treated with cast immobilization, with the removed cast in the preceding seven days.
* Approval from the orthopedic specialist to weight-bear as tolerated or partial weight-bear. -- Their ages will be between the age of 18 to 50 years of age.
* Participants having no concurrent injuries or pathology, such as neurological injury or other fractures.

Exclusion Criteria:

* Patients with surgical fixation,
* Fracture malunion or nonunion,
* Syndesmosis injury, or any standard contraindication to manual physical therapy.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-08-25 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
1. EMG assessment of muscle activity: | 2 momths
  Electromyogram (EMG) is the recording of the muscle activity and in this study EMG will be recorded from the tibialis anterior (TA) and the triceps surae muscle groups: medial gastrocnemius (MG), lateral gastrocnemius (LG) and soleus (SOL). Myomonitor 4 (Delsys, Boston) EMG data acquisition system was used. This has a gain of 1000, CMRR of 92 dB and bandwidth of 20-450 Hz, and 12 dB/octave roll-off. The sampling rate was 1000 Hz with a resolution of 16 bits/sample. Delsys single-channel active differential silver bar (10 mm x 1 mm) were used to record EMG. These will be embedded preamplifiers and fixed inter-electrode distance of 10 mm.

SECONDARY OUTCOMES:
Dynamic Plantar Pressure | 2 months.
  Dynamic plantar pressure was recorded using a single BTS P-WALK pressure platform (BTS Bioengineering S.p.A. Italy), with dimensions 640 mm _ 740 mm _ 8 mm and an acquisition frequency of 250 Hz. Data transmission to the computer is via USB2, where specific software (BTS G-Studio) processes the information received. The software itself identifies each step performed, and in the processing, the researchers themselves (M.F.-G. and D.S.-G.) take care of eliminating incorrect or incomplete steps .
  For data collection, the pressure platform was placed in the intermediate part (4 m) of the walkway. In this way, for step standardization, we ensured that at least three steps were taken before stepping on the plate. Five steps were collected with each limb during a continuous gait cycle. The variables recorded using the pressure platform were: weight-normalised peak plantar pressure (PPP) (kPa)-peak pressure recorded from the total number of steps taken during the gait.
Berg Balance Scale (BBS): | 2 months.
  The Berg balance scale includes 14 items with scores from 0 to 4. A score of 0 represents the inability to do the task, while a score of 4 represents the ability to do the task completely, according to the assigned criteria, with 56 indicates the total score. Items range from tasks of simple mobility (e.g. transfers, standing unsupported, sit-to-stand) to tasks with greater difficulty.
Ankle Joint Dorsiflexion and Planterflexion Range (ROM): | 2 months.
  Passive ankle-dorsiflexion and planterflexion ROM will be measured in 2 positions (extended knee and flexed knee) using a standard manual goniometer. For the extended-knee assessment, Patients will be seated on a treatment table with the knees fully extended (0°) and the feet hanging off the end of the table. For the flexed-knee assessment, they will be seated with the popliteal space at the edge of the table and the knees in 90° of flexion. For each ROM measurement, the participant will be completely relaxed; the investigator will passively moved the ankle into dorsiflexion and planterflexion from a neutral starting position (ie, 90° angle between shank and foot segments) until a firm end feel will be elicited. The axis of the goniometer will be centered over the lateral malleolus and the arms will be aligned with the fibular shaft and the head of the fifth metatarsal.
Pain Assessment. | 2 months.
  By numerical rating scale: The 11-point numerical pain rating scale was used in this study to indicate the intensity pain. It is composed of a numeric segmented horizontal line ranging from 0 which represents "no pain" and 10 which represents "worst imaginable pain." The scale was explained to each participant before using to ensure efficiency. Each participant was instructed to choose a numerical value (from 0 to 10 integers) that best describes the intensity of his pain in the preceding 24 hours.

CONTACTS AND LOCATIONS:
Locations (1):
- Hadaya Mosaad Eladl, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared after 6 months of publication.
Supporting Information: Study Protocol, ICF
Time Frame: 6 Months after publication.
Access Criteria: The study protocol and Informed Consent form will be shared after 6 months of publication.

REFERENCES:
- [Derived] Eladl HM, Elsherbini DMA, Elshorbagy RT, Ibrahim AM, El-Sherbiny M, Ibrahim SEAE, Elfayoumi GIF, Aboonq MS, Elbastawisy YM, Salama MEM, Allam NM. Efficacy of adding mobilization and balance exercises to a home-based exercise program in patients with ankle disability: a randomized controlled trial. Front Med (Lausanne). 2025 Feb 19;12:1512587. doi: 10.3389/fmed.2025.1512587. eCollection 2025. PMID 40046922